CLINICAL TRIAL: NCT06755515
Title: A Phase Ⅱ/Ⅲ Randomized, Double-Blind, Placebo-Controlled Trial of Rulonilimab Plus Chemotherapy± Bevacizumab for the First-Line Treatment of Persistent, Recurrent or Metastatic Cervical Cancer
Brief Title: A Phase Ⅱ/Ⅲ Study of Rulonilimab Plus Chemotherapy± Bevacizumab for the First-Line Treatment of Persistent, Recurrent or Metastatic Cervical Cancer
Status: Enrolling by invitation | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Shandong New Time Pharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NTP-F520-502
Record Dates: First submitted 2024-12-24; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-12

CONDITIONS: Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Cisplatin; Carboplatin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rulonilimab plus cisplatin/carboplatin + paclitaxel ± bevacizumab (Experimental)
  Interventions: Drug: Rulonilimab; Drug: cisplatin/carboplatin + paclitaxel ± bevacizumab
- Placebo plus cisplatin/carboplatin + paclitaxel ± bevacizumab (Placebo Comparator)
  Interventions: Drug: Placebo; Drug: cisplatin/carboplatin + paclitaxel ± bevacizumab

INTERVENTIONS:
Drug: Rulonilimab — Drug: Rulonilimab Description: iv, 200mg every 3 weeks, for up to 2 years until disease progression, intolerable toxic reactions, or termination of treatment for other reasons.
  Drug: Bevacizumab Description: iv, 15mg/kg every 3 weeks, for up to 2 years until disease progression, intolerable toxic reactions, or termination of treatment for other reasons.
  Drug: Cisplatin Description: iv, 50mg/m^2 every 3 weeks, for up to 6 cycles. Drug: Carboplatin Description: iv, AUC 4~6 every 3 weeks, for up to 6 cycles. Drug: Paclitaxel Description: iv, 175mg/m^2 every 3 weeks, for up to 6 cycles.
  Arms: Rulonilimab plus cisplatin/carboplatin + paclitaxel ± bevacizumab
Drug: Placebo — Drug: placebo Description: iv, every 3 weeks, for up to 2 years until disease progression, intolerable toxic reactions, or termination of treatment for other reasons.
  Drug: Bevacizumab Description: iv, 15mg/kg every 3 weeks, for up to 2 years until disease progression, intolerable toxic reactions, or termination of treatment for other reasons.
  Drug: Cisplatin Description: iv, 50mg/m^2 every 3 weeks, for up to 6 cycles. Drug: Carboplatin Description: iv, AUC 4~6 every 3 weeks, for up to 6 cycles. Drug: Paclitaxel Description: iv, 175mg/m^2 every 3 weeks, for up to 6 cycles.
  Arms: Placebo plus cisplatin/carboplatin + paclitaxel ± bevacizumab
Drug: cisplatin/carboplatin + paclitaxel ± bevacizumab — cisplatin/carboplatin + paclitaxel ± bevacizumab

SUMMARY:
This study was an randomized, double-Blind, placebo-controlled, multicenter Phase II/III study.

DETAILED DESCRIPTION:
The trial was divided into screening period, treatment period and follow-up period. Participants entered the screening period after signing informed consent and met the inclusion criteria. Subjects who did not meet the exclusion criteria were treated with Rulonilimab/placebo plus chemotherapy ± bevacizumab, intravenously, at target dose every 3 weeks until disease progression or intolerable toxicity or withdrawal for other reasons, for a maximum of 2 years.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged 18 years and above;
2. Patients with advanced ([FIGO] stage IVB) cervical cancer, patients with persistent, recurrent or metastatic cervical cancer that progresses confirmed by histopathology or cytology, and the following conditions must be met:

   Programmed Cell Death Ligand 1 (PD-L1) positive expression defined by Combined Positive Score (CPS) ≥1; The histopathology types include squamous cell carcinoma, adenocarcinoma, or adenosquamous cell carcinoma; Not amenable to curative surgery or concurrent chemoradiotherapy; No prior systemic therapy for advanced, persistent, recurrent or metastatic disease; Patients who had previously received first-line platinum-containing adjuvant or neoadjuvant chemotherapy/radical concurrent chemoradiotherapy and whose time from the last chemotherapy to disease progression was > 6 months were eligible for inclusion.
3. According to RECIST1.1 criteria, subjects must have at least one measurable target lesion examined by Imaging tests (including Not to receive radiation therapy or other locoregional therapy unless the lesion PD or has tumor activity by biopsy-confirmed);
4. Those with 0-1 scores on the American Eastern Oncology Collaboration Group (ECOG) scale
5. Expected survival ≥3 months;
6. Those who agree to provide archived tumor tissue samples or before randomized within 3 years or fresh tissue samples;
7. The function of vital organs meets the following requirements (drugs with blood components and cell growth factors are not allowed to be used within 2 weeks before the first administration) :

   Blood routine: Absolute neutrophil count ≥1.5×109/L; Platelet ≥75×109/L; Hemoglobin ≥90g/L; Liver function: TBIL≤1.5×ULN, ALT and AST≤2.5×ULN; If liver metastasis was present, TBIL≤3×ULN, ALT and AST≤5×ULN; Renal function: serum creatinine (Cr) ≤1.5×ULN a creatinine clearance (CrCl) ≥ 50 mL/min if Cr>1.5×ULN; Coagulation function: International Normalized ratio (INR) ≤1.5×ULN and activated partial thromboplastin time (APTT) ≤1.5×ULN.

   Thyroid function: Thyroid stimulating hormone (TSH) in the normal range; If TSH is abnormal, free triiodothyronine (FT3) and free thyroxine (FT4) must be normal or abnormal without clinical significance.
8. Willingness to participate in the clinical trial; completely understanding and knowing about the study and signing the ICF; willingness and capability to comply with the requirements of the study.

Exclusion Criteria:

1. Patients with pathological tissue types of mucinous adenocarcinoma, gastric adenocarcinoma, clear cell adenocarcinoma, mesonephric tubular adenocarcinoma and other special types of adenocarcinoma；
2. Those who previously treated with T-cell co-stimulation, Antiangiogenic drugs (bevacizumab), immune checkpoint inhibitor (anti-PD-1, anti-PD-L1, anti-PD-L2, or anti-CTLA-4 antibodies), Targeting immune co-stimulatory factors drug (ICOS, CD40, CD137, GITR, OX40 antibodies);
3. Those who have received anti-tumor treatment within 4 weeks before the first dose or within 5 half-lives of the drug (whichever is shorter);
4. Immunosuppressive, systemic hormone therapy within 2 weeks prior to initial administration for immunosuppressive purposes (daily dose equivalent to prednisone>10mg of systemic corticosteroid);
5. The toxicity of previous anti-tumor therapy did not return to CTCAE V5.0 ≤ grade 1 (except hair loss);
6. A history of other malignancies within the last 5 years, except locally curable cancers (limited to Radical melanoma, basal cell or squamous cell skin cancer, superficial bladder cancer, or carcinoma in situ of the breast);
7. Patients with primary central nervous system (CNS) malignancies, CNS metastases that have failed local treatment, and carcinomatous meningitis; the following conditions can be included (regular imaging examinations of the disease site): a. No progressive CNS symptoms caused by brain metastases, no need for steroid hormone treatment, and the lesion is less than 1.5 cm; b. Stable for ≥4 weeks after adequate treatment and neurological symptoms (excluding residual signs or symptoms) have returned to baseline levels for >2 weeks before the first dose;
8. Patients with uncontrollable pleural effusion, pericardial effusion or peritoneal effusion that requires repeated drainage (more than once a month) (can be enrolled after stable treatment for more than 1 month);
9. Patients with a history of organ transplantation or allogeneic bone marrow transplantation; or autologous stem cell transplantation within 3 months before the first dose;
10. Patients who have undergone major surgery or have not yet recovered from surgery within 4 weeks before the first dose (except for diagnostic surgery);
11. Physical examination or laboratory test findings:

    Hepatitis B: HBsAg positive and/or HBcAb positive, and HBV-DNA>500IU/mL or 2500 copies/mL; Hepatitis C: HCV antibody positive, and HCV-RNA positive or above the upper limit of normal value; Human immunodeficiency virus antibody (Anti-HIV) positive; Active Treponema pallidum infection;
12. Patients with thrombosis who need treatment in the acute stage;
13. Those who have uncontrolled or severe cardiovascular disease, such as New York Heart Association (NYHA) Class II or above congestive heart failure or LVEF<50%, unstable angina, myocardial infarction and other cardiovascular disease within 6 months before the first dose; Poorly controlled arrhythmias; Difficult to control hypertension (systolic blood pressure ≥160mmHg and/or diastolic blood pressure ≥100mmHg after drug therapy);
14. Patients with the following medical histories, including but not limited to active autoimmune diseases, active infections (such as active tuberculosis), severe mental illness, severe endocrine diseases (such as type 1 diabetes, type 2 diabetes that cannot be controlled by drugs), etc.;
15. have been treated with any other investigational drug/device within 4 weeks prior to initial dosing;
16. Those who have a history of drug abuse or alcoholism within 6 months before the first dose;
17. Those with a history of severe allergies, known subjects to have been allergic to macromolecular protein preparations/monoclonal antibodies and any components of the experimental drugs;
18. Those who have received live or attenuated live vaccines within 4 weeks before the first dose or are scheduled to receive live or attenuated live vaccines during the study;
19. Pregnant or lactating women, and female subjects of childbearing age who do not agree to use medically recognized effective contraceptive measures (such as intrauterine devices or condoms) during the study and within 6 months after the last trial drug treatment;
20. Those who were judged not suitable for inclusion by the researchers.
21. The following conditions are only applicable to those who are excluded from the use of bevacizumab:

    1. Within 3 months before the first dose, there is clinically significant hematuria, hematemesis or hemoptysis (>2.5mL red blood), or other history of obvious bleeding (such as pulmonary hemorrhage);
    2. Patients who are receiving thrombolytic/anticoagulant therapy, or need to continue to receive thrombolytic/anticoagulant therapy during the study (prophylactic use of low-dose aspirin is allowed);
    3. Patients with unhealed, poorly healed wounds or untreated fractures;
    4. Patients with evidence of gastrointestinal perforation, fistula, intra-abdominal abscess, and free gas in the abdominal cavity within 6 months before the first dose;
    5. Subjects with urine protein>1+ undergo 24-hour urine protein quantification, and urine protein ≥1g/24 hours;
    6. Patients with reversible posterior encephalopathy syndrome (PRES) or reversible posterior leukoencephalopathy syndrome (RPLS).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2024-09-26 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Objective tumor response rate (ORR) assessed by RECIST1.1 | up to 2 years
  Defined as the proportion of subjects who achieves a best overall response of CR or PR based on RECIST1.1
Progression Free Survival (PFS) assessed by RECIST1.1 | up to 2 years
  Defined as the time from the date of randomization to the date of progressive disease (PD) or death, whichever occurs first.
Overall Survival (OS) | up to 2 years
  Defined as the time from the date of randomization to the date of death due to any Defined as the time from the date of randomization to the date of death due to any reason

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | up to 2 years
  Defined as the proportion of subjects' response of CR, PR, or SD based onRECIST1.1
Duration of Response (DOR) | up to 2 years
  Defined as the time from the date that CR or PR are first occurred to the date of objective disease progression or death, whichever occurs first
Time to Response (TTR) | up to 2 years
  Defined as the time from the date of randomization to the date when the response criteria are first met, based on RECIST1.1

OTHER OUTCOMES:
The Incidence and Severity of adverse events (AEs) and serious adverse events (SAEs) | up to 2 years
  Number of participants with an AE or SAE
Healthy related quality of life (HRQoL) | up to 2 years
  EORTC QLQ-C30 will be used

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong New Time Pharmaceutical Co., LTD, Linyi, Shandong, China